CLINICAL TRIAL: NCT02971293
Title: A Phase IIa, Randomised, Multi-Centre, Double-Blind, Placebo-Controlled, 3 Periods, Crossover Study to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of Inhaled AZD8871 Administered Once Daily for 2 Weeks in Patients With Moderate to Severe COPD.
Brief Title: Efficacy, Pharmacokinetics (PK), Safety and Tolerability Study of Inhaled AZD8871
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D6640C00004
Record Dates: First submitted 2016-10-28; First posted 2016-11-22 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
Keywords: AZD8871; long-acting muscarinic antagonist (LAMA); long-acting β2-agonist (LABA); inhaled long-acting bronchodilator; pharmacokinetics; safety; tolerability; efficacy; Phase IIa; Muscarinic receptor antagonist β2 adrenoceptor agonist (MABA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD-8871

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZD8871 100 µg (Experimental): The subjects will receive AZD8871 100 µg once daily, by dry powder inhaler (DPI) device. The treatment will be administered via single dose DPI that is an adaptation of the multi-dose Genuair™ used in approved inhalation products.
  Interventions: Drug: AZD8871 100 µg
- Placebo (Placebo Comparator): The placebo will be administered via single dose DPI that is an adaptation of the commercially available Genuair® with a smaller internal volume to enable delivery of single doses. To maintain blinding, each patient will receive one inhaled dose from placebo DPI provided to him/her on each day of the treatment period.
  Interventions: Drug: Placebo
- AZD8871 600 µg (Experimental): The subjects will receive AZD8871 600 µg once daily by DPI device via single dose DPI that is an adaptation of the multi-dose Genuair™ used in approved inhalation products.
  Interventions: Drug: AZD8871 600 µg

INTERVENTIONS:
Drug: AZD8871 100 µg — The subjects will receive one dose of AZD8871 100 µg single dose DPI.
  Arms: AZD8871 100 µg
Drug: AZD8871 600 µg — The subjects will receive AZD8871, 600 µg single dose DPI.
  Arms: AZD8871 600 µg
Drug: Placebo — The subject will receive Placebo single dose DPI.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the effects of AZD8871 in patients with COPD. Adult male or female patients with moderate to severe COPD, who agree to be in this study, will receive 3 treatments, i.e. 2 different doses of AZD8871 and placebo (dummy medication containing no drug) at once a day for 2 weeks, in a random order. To make the comparison between AZD8871 and placebo as fair as possible, this study is "double blinded." This means that neither patient nor the study doctor will know in which order the 3 treatments will be given. This study will include patients who are between 40 and 80 years of age. In total there will be 42 patients participating in this study at two study centers in the United Kingdom and Germany. The study will have a total of 12 visits for each patient spanning for a period of 4 to 6 months. The study is anticipated to run for approximately 8 months and should not exceed 10 months.

DETAILED DESCRIPTION:
This is a proof-of-concept, randomised, double-blind, placebo-controlled, 3-way, complete crossover William's design, multiple dose study to investigate the efficacy, PK, safety, and tolerability of 2 dose levels of AZD8871 and placebo, administered using a dry powder inhaler (DPI) device once daily, for 2 weeks, in patients with moderate to severe COPD. AZD8871 is a new chemical entity with the combined properties of a LAMA and a LABA in a single molecule. AZD8871 is being developed as an inhaled long-acting bronchodilator for the maintenance treatment of COPD.

The objective of the study is to assess the efficacy, safety and PK of AZD8871 after a 14-day treatment period at 2 different doses in patients with moderate to severe COPD. The target population includes male and female (non-childbearing potential) adult patients with clinical diagnosis of moderate to severe COPD. The crossover design has been chosen to avoid inter-patient variability and optimize sample size. By randomly assigning treatment sequence, differences in baseline characteristics of the treatment groups will be minimised. The inclusion of a placebo arm is considered the most reliable method to minimise patient and Investigator bias. The proposed dose levels of AZD8871 in this study are 100 and 600 µg of AZD8871 given by inhalation once daily for 14 days through a single dose DPI. Doses have been selected based on the safety, tolerability, PK and pharmacodynamics (PD) information generated in previous clinical trials with AZD8871. The wash-out period proposed for this current study is a minimum of 28 days and up to 35 days in order to avoid any carry over effect between periods. The broad dose range selected (6 fold range from 100 to 600 µg) has been chosen to span the likely therapeutic dose and facilitate the dose selection for future studies. Considering the expected efficacy in patients with COPD and the available data to date, it is anticipated the benefits will outweigh the risks and support the continued investigation of AZD8871 in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who provided of informed consent prior to any study-specific procedures
2. Male or female 40 to 80 years of age (both inclusive) at Screening (Visit 1). A female is eligible to enter and participate in the study if she is of non-childbearing potential.

   Note: A female is considered to be of non-childbearing potential if she meets one of the following criteria:
   * Permanently or surgically sterilised, including hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy
   * Post-menopausal; aged <50 years and amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range of the local laboratory.
   * Post-menopausal; aged ≥50 years and amenorrhoeic for 12 months or more, following cessation of all exogenous hormonal treatments.
3. Male patient should use a condom and spermicide to prevent pregnancy and drug exposure of a partner, regardless of the gender or childbearing potential of the partner from the day of the first administration of the investigational product (IP) until 3 months after the last administration of the IP.
4. COPD Diagnosis: Patient with an established clinical history of COPD for more than 1 year at Screening, according to the Global Initiative for Chronic Obstructive Lung Disease 2016 COPD guidelines.
5. Tobacco Use: Patient is a current or former smoker with a history of ≥10 pack-years of cigarette smoking. A former smoker is defined as one who has stopped smoking for at least 6 months prior to Screening.
6. Patient with post-bronchodilator FEV1/FVC (Forced vital capacity) ratio <70% based on the value reached after inhalation of salbutamol (400 µg) at Visit 2. If criterion is not met, the test can be repeated at the latest, up to Day 14.
7. Patient with post-bronchodilator FEV1 that must be ≥40% and <80% predicted normal value and must also be >750 mL at Visit 2. If criterion is not met, the test can be repeated at the latest, up to Day 14.
8. Patient who fulfils reversibility criteria to salbutamol at Visit 2. Reversibility is defined as ≥12% and ≥200 mL increase in FEV1 after inhalation of 4 puffs of salbutamol. (400 µg). If criterion is not met, the test can be repeated at the latest, up to Day 14.
9. Patient is willing and, in the opinion of the Investigator, able to change current COPD therapy as required by the protocol and willing to use ipratropium Four times a day (if needed, during run-in and wash-out periods) with or without Inhaled corticosteroid for maintenance therapy of COPD and as needed rescue salbutamol from Visit 1 up Visit 11.
10. Patient is free from any clinically active disease other than COPD that may impact study outcome, as determined by medical history, physical examination, laboratory testing, and 12-lead ECG findings, at Screening.
11. Patient is willing to remain at the study centre as required per protocol to complete all visit assessments.
12. Patient with body mass index (BMI) <40 kg/m2 at the time of screening.

Exclusion Criteria:

1. Patient previously enrolled in the present study.
2. Patient has significant diseases other than COPD, ie, disease or condition or an abnormality in laboratory, ECG, medical history or physical examination which, in the opinion of the Investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patient'spatient's ability to participate in the study.
3. Childbearing potential female, pregnant or lactating.
4. Patient who, in the opinion of the Investigator, has a current diagnosis of asthma.
5. Patient has alpha-1 antitrypsin deficiency as the cause of COPD.
6. Patient has other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnoea. Allergic rhinitis is not exclusionary.
7. Lung surgery for volume reduction or lung transplantation: Patient has undergone lung volume reduction surgery, lobectomy, or bronchoscopic lung volume reduction (endobronchial blockers, airway bypass, endobronchial valves, thermal vapour ablation, biological sealants, massive pulmonary embolism and airway implants) within 1 year of Screening (Visit 1).
8. Patient is using nocturnal positive pressure (eg, continuous positive airway pressure or bi level positive airway pressure). Patient is using any non-invasive positive pressure ventilation device.

   Note: A patient using continuous positive airway pressure or bi level positive airway pressure for Sleep Apnoea Syndrome is allowed in the study.
9. Patient has been hospitalised due to poorly controlled COPD within 3 months of Screening.
10. Patient has acute worsening of COPD that requires treatment with corticosteroids or antibiotics in the 6 week interval prior to Screening (Visit 1), or during the Screening Period (between Visits 1 and 3).
11. Patient has had lower respiratory tract infections that required antibiotics within 6 weeks prior to Screening.
12. Patient cannot perform acceptable spirometry, ie, meet American Thoracic Society (ATS)/European Respiratory Society (ERS) acceptability criteria.
13. Patient has changed their smoking status (ie, start or stop smoking) or initiation of a smoking cessation program within 6 weeks prior to Screening.
14. Patient has participated in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening or who will enter the acute phase of a pulmonary rehabilitation program during the study. A patient in the maintenance phase of a pulmonary rehabilitation program is not to be excluded.
15. Cardiac disease: Subject with significant cardiovascular disease cardiovascular instability. Patient with heart rate <50 beats per minute. Patient has clinically significant uncontrolled hypertension as assessed by the investigator.
16. Neurological: Patient with seizures or history of seizures requiring anticonvulsants within 12 months prior to Screening. Patient is taking selective serotonin reuptake inhibitors or serotonin--norepinephrine reuptake inhibitors whose dose has not been stable for at least 4 weeks prior to Screening, or exceeds the maximum recommended dose.
17. Renal: Patient with symptomatic bladder neck obstruction, acute urinary retention or symptomatic non-stable prostate hypertrophy. 35.23. Patient with a serum potassium value <3.5 mmol/L at Screening and on repeat testing. Note: however potassium replacement and rescreening is allowed if serum potassium concentration was < 3.5mmol/l at screening.
18. Others:

    * Any laboratory abnormality or suspicion of any clinically relevant disease or disorder (on history or examination), including uncontrolled hypertension or uncontrolled diabetes, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study, or any other safety concerns in the opinion of the Investigator.
    * History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin
    * Patient with known narrow-angle glaucoma.
    * Patient has a history of hypersensitivity to β2-agonists, muscarinic anticholinergics or lactose/milk protein. Lactose intolerance is not an exclusion criterion.
    * The patient has a known or suspected history of alcohol or drug of abuse within the past 2-year period years or consuming more than 14 (female subjects) or 21 (male subjects) units of alcohol a week, or shows positive for drugs of abuse and alcohol tests at screening and prior to randomization.
    * Patient who, in the opinion of the Investigator, would be unable to abstain from protocol-defined prohibited medications during the study.
    * Patient who received a live attenuated vaccination within 30 days prior to Screening.
    * Patient involved in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
    * Patient treated with investigational drug or device in another clinical trial within the last 30 days or five half-lives (whichever is longer) prior to Screening.
    * Patient who donated or lost >500 mL of blood and plasma within the previous 3 months prior to screening.
    * Patient is unlikely to co-operate with the requirements of the study, instructions of the Principal Investigator., or have e-dairy completion rate of < 70% during the run in period.
    * Patient with known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C infection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Prof, Principal Investigator — Medicines Evaluation Unit, Manchester, United Kingdom; Rainard Fuhr, Dr, Principal Investigator — PAREXEL International GmbH EPCU Berlin
Locations (2):
- Research Site, Berlin, Germany
- Research Site, Manchester, United Kingdom

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4121&filename=AZD8871%20D6640C00006%20Clinical%20Study%20Protocol%20(CSP)_redacted.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4121&filename=azd8871-d6640c00004-redacted-sap-ed-1-3.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at two centres, one each in Germany and the UK. The first patient was enrolled in December 2016 and the last patient last visit was in August 2017.
Pre-assignment Details: A total of 103 patients were screened; 42 patients were eligible to participate and were randomised.
Groups:
- All Participants: All subjects received AZD8871 100 µg, AZD8871 600 µg or placebo, once daily by DPI device via single dose DPI that is an adaptation of the multi-dose Genuair™ used in approved inhalation products.
  Each subject was randomized to one of three sequences in a 3-way, complete crossover William's design, and received all 3 treatments in turn, in three 14-day treatment periods, each (except the last one) followed by a wash-out period of 28-35 days.
Period: Overall Study
Arm/Group | All Participants
Started (3-way, complete crossover. Each patient received all 3 treatments in turn; randomised sequence.) | 42
Completed | 31
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Safety analysis set: Includes all randomised participants who received at least one dose of investigational product.
Groups:
- Overall Study Population: Full analysis set: All randomised participants who received at least one dose of investigational product.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (6.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change in trough FEV1 on Day 15
Time Frame: On Day 15
Population: Full analysis set (FAS): all randomised patients who received at least one dose of the IP, irrespective of their protocol adherence and continued participation in the study.
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- AZD8871 100 µg: The subjects received AZD8871 100 µg once daily by DPI device via single dose DPI that is an adaptation of the multi-dose Genuair™ used in approved inhalation products.
- AZD8871 600 µg: The subjects received AZD8871 600 µg once daily by DPI device via single dose DPI that is an adaptation of the multi-dose Genuair™ used in approved inhalation products.
- Placebo: The placebo was administered via single dose DPI that is an adaptation of the commercially available Genuair® with a smaller internal volume to enable delivery of single doses. To maintain blinding, each patient received one inhaled dose from placebo DPI provided to him/her on each day of the treatment period.
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.168 (0.037) | 0.267 (0.035) | 0.007 (0.036)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; Fixed effects: treatment, sequence, period. Random effect for patient nested within sequence. Continuous covariate: baseline
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.020, ANCOVA; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Observed Maximum Plasma (Cmax) of AZD8871 and Its Metabolites (Single Dose)
Description: Observed maximum concentration, taken directly from the individual concentration-time curve, on Day 1 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1.
Population: Pharmacokinetic analysis set: defined as all patients in the safety analysis set who received at least 1 dose of AZD8871 (100 μg or 600 μg), had at least 1 evaluable parameter out of Cmax, AUC or AUClast for AZD8871, and were assumed not to be affected by factors such as protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg/mL
  AZD8871 | 61.05 (47.47) | 290.8 (36.30) |
  LAS191861 | 7.796 (38.67) | 33.87 (33.05) |
  LAS34850 | 187.7 (55.41) | 1016 (50.72) |

3. Secondary Outcome: Observed Maximum Plasma (Cmax) of AZD8871 and Its Metabolites (Multiple Doses, Day 14)
Description: Observed maximum concentration, taken directly from the individual concentration-time curve, on Day 14 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg/mL
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 72.52 (45.69) | 381.8 (36.09) |
  LAS191861: number analyzed (Participants) | 16 | 17 | 0
  LAS191861 | 11.89 (39.41) | 63.17 (38.23) |
  LAS34850: number analyzed (Participants) | 16 | 17 | 0
  LAS34850 | 221.4 (69.96) | 1152 (55.11) |

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of AZD8871 and Its Metabolites (Single Dose)
Description: Time to reach maximum concentration taken directly from the individual concentration-time curve on Day 1 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1.
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
h
  AZD8871 | 0.93 [0.42 to 2.00] | 1.46 [0.48 to 2.03] |
  LAS191861 | 1.92 [0.93 to 4.83] | 2.02 [1.00 to 4.03] |
  LAS34850 | 3.94 [1.92 to 6.00] | 3.98 [3.92 to 6.03] |

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of AZD8871 and Its Metabolites (Multiple Doses, Day 14)
Description: Time to reach maximum concentration taken directly from the individual concentration-time curve on Day 14 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 14.
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
h
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 0.93 [0.42 to 1.00] | 1.00 [0.50 to 2.22] |
  LAS191861: number analyzed (Participants) | 16 | 17 | 0
  LAS191861 | 1.96 [0.98 to 3.95] | 2.00 [0.98 to 3.98] |
  LAS34850: number analyzed (Participants) | 16 | 17 | 0
  LAS34850 | 3.92 [0.00 to 4.00] | 4.02 [3.90 to 6.05] |

6. Secondary Outcome: AUClast of AZD8871 and Its Metabolites (Single Dose)
Description: Area under the plasma concentration-curve from time zero to the last quantifiable time point (24 hours post-dose) calculated on Day 1 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg*h/mL
  AZD8871 | 301.0 (54.52) | 1777 (40.93) |
  LAS191861 | 60.06 (94.87) | 358.5 (32.60) |
  LAS34850: number analyzed (Participants) | 14 | 18 | 0
  LAS34850 | 1414 (69.31) | 9299 (53.88) |

7. Secondary Outcome: AUClast of AZD8871 and Its Metabolites (Multiple Doses, Day 14)
Description: Area under the plasma concentration-curve from time zero to the last quantifiable time point (24 hours post-dose) calculated on Day 14 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg*h/mL
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 539.2 (51.23) | 3156 (42.51) |
  LAS191861: number analyzed (Participants) | 16 | 17 | 0
  LAS191861 | 160.2 (64.39) | 935.9 (46.56) |
  LAS34850: number analyzed (Participants) | 15 | 17 | 0
  LAS34850 | 1964 (93.81) | 13050 (52.49) |

8. Secondary Outcome: AUC0-24 of AZD8871 and Its Metabolites (Single Dose)
Description: Area under the plasma concentration-curve from time zero to 24 hours post-dose calculated on Day 1 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg*h/mL
  AZD8871: number analyzed (Participants) | 14 | 18 | 0
  AZD8871 | 326.1 (49.18) | 1776 (40.95) |
  LAS191861: number analyzed (Participants) | 7 | 18 | 0
  LAS191861 | 135.6 (25.79) | 358.1 (32.56) |
  LAS34850: number analyzed (Participants) | 1 | 15 | 0
  LAS34850 | 0 (0) | 10440 (49.47) |

9. Secondary Outcome: AUC0-24 of AZD8871 and Its Metabolites (Multiple Doses, Day 14)
Description: Area under the plasma concentration-curve from time zero to 24 hours post-dose calculated on Day 14 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg*h/mL
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 538.4 (51.16) | 3152 (42.53) |
  LAS191861: number analyzed (Participants) | 15 | 17 | 0
  LAS191861 | 179.4 (38.81) | 933.8 (46.65) |
  LAS34850: number analyzed (Participants) | 7 | 17 | 0
  LAS34850 | 3281 (66.13) | 13030 (52.51) |

10. Secondary Outcome: Accumulation Ratio for Cmax (RacCmax) of AZD8871 and Its Metabolites (Day 14)
Description: Accumulation ratio for Cmax estimated as (Cmax on Day 14 / Cmax on Day 1) in each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 14.
Population: as for outcome 2
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg/mL
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 1.263 [0.765 to 2.30] | 1.385 [0.700 to 1.90] |
  LAS191861: number analyzed (Participants) | 16 | 17 | 0
  LAS191861 | 1.594 [0.946 to 2.86] | 1.968 [0.929 to 2.74] |
  LAS34850: number analyzed (Participants) | 16 | 17 | 0
  LAS34850 | 1.257 [0.757 to 3.388] | 1.133 [0.545 to 1.64] |

11. Secondary Outcome: Accumulation Ratio for AUC0-24 (RacAUC[0-24]) of AZD8871 and Its Metabolites (Day 14)
Description: Accumulation ratio for AUC0-24 estimated as AUC0-24 on Day 14 / AUC0-24 on Day 1 in each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 1 and Day 14.
Population: as for outcome 2
Measure: Mean (Full Range); unit: pg*h/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg*h/mL
  AZD8871: number analyzed (Participants) | 14 | 17 | 0
  AZD8871 | 1.893 [1.06 to 3.86] | 1.878 [1.09 to 2.87] |
  LAS191861: number analyzed (Participants) | 7 | 17 | 0
  LAS191861 | 1.576 [1.10 to 2.44] | 2.721 [1.41 to 3.55] |
  LAS34850: number analyzed (Participants) | 1 | 15 | 0
  LAS34850 | 1.24 [1.24 to 1.24] | 1.326 [0.713 to 1.77] |

12. Secondary Outcome: Cavg of AZD8871 and Its Metabolites During a Dosing Interval (Day 14)
Description: Average plasma concentration during a dosing interval calculated on Day 14 of each treatment period.
Time Frame: Pre-dose and 30 min, 1, 2, 4, 6, 8, 12, and 24 hours post-dose on Day 14.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 16 | 18 | 0
pg/mL
  AZD8871: number analyzed (Participants) | 16 | 17 | 0
  AZD8871 | 22.44 (51.13) | 131.4 (42.49) |
  LAS191861: number analyzed (Participants) | 15 | 17 | 0
  LAS191861 | 7.478 (38.81) | 38.94 (46.62) |
  LAS34850: number analyzed (Participants) | 7 | 17 | 0
  LAS34850 | 136.7 (66.11) | 543.3 (52.44) |

13. Secondary Outcome: Change From Baseline in Trough FEV1 at Day 1 (Single Dose)
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change in trough FEV1 on Day 1
Time Frame: on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.092 (0.029) | 0.161 (0.027) | 0.006 (0.028)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.011, ANCOVA; [statistical method as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Trough FEV1 at Day 8 (Pre-dose)
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change in trough FEV1 on Day 8 (pre-dose)
Time Frame: on Day 8 (pre-dose)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.180 (0.033) | 0.232 (0.030) | 0.032 (0.031)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.201, ANCOVA; [statistical method as in outcome 1, analysis 1]

15. Secondary Outcome: Change From Baseline in Trough FEV1 Over the Treatment Duration (Days 1-15)
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change in trough FEV1 over the treatment duration from Day 1 to Day 15
Time Frame: Days 1-15
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.146 (0.029) | 0.215 (0.027) | 0.016 (0.027)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; Fixed effect: treatment, sequence, period, treatment*day. Repeat factor: day. Random effect: patient nested in sequence. Continuous covar: baseline
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.020, ANCOVA; [statistical method as in outcome 15, analysis 1]

16. Secondary Outcome: Change From Baseline in Peak FEV1 at Day 1 (Single Dose)
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change in Peak FEV1
Time Frame: on Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.376 (0.026) | 0.469 (0.025) | 0.076 (0.025)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]

17. Secondary Outcome: Change From Baseline in Peak FEV1 at Day 8
Description: as for outcome 16
Time Frame: on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.486 (0.040) | 0.556 (0.037) | 0.136 (0.038)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.092, ANCOVA; [statistical method as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in Peak FEV1 at Day 14
Description: as for outcome 16
Time Frame: on Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.476 (0.037) | 0.522 (0.035) | 0.095 (0.036)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.279, ANCOVA; [statistical method as in outcome 1, analysis 1]

19. Secondary Outcome: Change From Baseline in Peak FEV1 Over the Treatment Duration (Days 1-15)
Description: as for outcome 16
Time Frame: over the treatment duration (Days 1-15)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
L | 0.438 (0.028) | 0.511 (0.027) | 0.102 (0.028)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 15, analysis 1]

20. Secondary Outcome: Change From Baseline in BCSS Questionnaire Total Score From Day 1 to Day 8 Post-treatment
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD was assessed by measuring the change from baseline in Total score of the Breathlessness, Cough Sputum Scale (BCSS) questionnaire.
  The BCSS questionnaire is a 3-item patient-reported outcome measure. On a daily basis, patients rated 3 symptoms (breathlessness, cough and sputum) on a 5-point Likert scale (range 0-4, high scores indicating higher severity). The BCSS questionnaire Total Score is the sum of the 3 symptom scores, ranging from 0-12 (lowest-highest severity).
Time Frame: From Day 1 to Day 8 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.416 (0.216) | -0.920 (0.198) | -0.071 (0.205)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.205, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.060, ANCOVA; [statistical method as in outcome 1, analysis 1]

21. Secondary Outcome: Change From Baseline in BCSS Questionnaire Total Score From Day 9 to Day 14 Post-treatment
Description: as for outcome 20
Time Frame: From Day 9 to Day 14 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.491 (0.237) | -1.191 (0.219) | -0.030 (0.226)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.111, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.015, ANCOVA; [statistical method as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Cough Individual Domain Score From Day 1 to Day 8 Post-treatment
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD will be assessed by measuring the change from baseline in Breathlessness, Cough Sputum Scale (BCSS) questionnaire cough individual domain scores.
  On a daily basis, patients rated cough symptoms on a 5-point Likert scale (range 0-4, high scores indicating higher severity).
Time Frame: From Day 1 to Day 8 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.186 (0.091) | -0.287 (0.084) | -0.134 (0.087)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.621, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p = 0.138, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.333, ANCOVA; [statistical method as in outcome 1, analysis 1]

23. Secondary Outcome: Change From Baseline in Cough Individual Domain Score From Day 9 to Day 14 Post-treatment
Description: as for outcome 22
Time Frame: From Day 9 to Day 14 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.160 (0.096) | -0.445 (0.088) | -0.123 (0.091)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.748, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.013, ANCOVA; [statistical method as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Breathlessness Individual Domain Score From Day 1 to Day 8 Post-treatment
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD will be assessed by measuring the change from baseline in Breathlessness, Cough Sputum Scale (BCSS) questionnaire breathlessness individual domain scores.
  On a daily basis, patients rated breathlessness symptoms on a 5-point Likert scale (range 0-4, high scores indicating higher severity).
Time Frame: From Day 1 to Day 8 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.122 (0.097) | -0.377 (0.089) | 0.099 (0.092)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.064, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.030, ANCOVA; [statistical method as in outcome 1, analysis 1]

25. Secondary Outcome: Change From Baseline in Breathlessness Individual Domain Score From Day 9 to Day 14 Post-treatment
Description: as for outcome 24
Time Frame: From Day 9 to Day 14 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.202 (0.108) | -0.453 (0.100) | 0.106 (0.103)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.018, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.047, ANCOVA; [statistical method as in outcome 1, analysis 1]

26. Secondary Outcome: Change From Baseline in Sputum Individual Domain Score From Day 1 to Day 8 Post-treatment
Description: The efficacy of inhaled AZD8871 in patients with moderate to severe COPD will be assessed by measuring the change from baseline in Breathlessness, Cough Sputum Scale (BCSS) questionnaire sputum individual domain scores.
  On a daily basis, patients rated sputum symptoms on a 5-point Likert scale (range 0-4, high scores indicating higher severity).
Time Frame: From Day 1 to Day 8 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.100 (0.070) | -0.255 (0.064) | -0.035 (0.066)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.477, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p = 0.014, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.084, ANCOVA; [statistical method as in outcome 1, analysis 1]

27. Secondary Outcome: Change From Baseline in Sputum Individual Domain Score From Day 9 to Day 14 Post-treatment
Description: as for outcome 26
Time Frame: From Day 9 to Day 14 post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
Number analyzed (Participants) | 34 | 39 | 36
Scores on a scale | -0.122 (0.078) | -0.297 (0.073) | -0.011 (0.075)
Statistical Analysis 1: Comparison: AZD8871 100 µg vs Placebo; Comparison of AZD8871 100 µg vs placebo; Test type: Superiority; p = 0.213, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: AZD8871 600 µg vs Placebo; Comparison of AZD8871 600 µg vs placebo; Test type: Superiority; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: AZD8871 100 µg vs AZD8871 600 µg; Comparison of AZD8871 600 µg vs AZD8871 100 µg; Test type: Superiority; p = 0.046, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From screening to Follow-up/early termination Visit, 28 to 35 days after the last administration of investigational product (IP)
Description: All reported AEs, date of onset, date of resolution, Investigator's assessment of severity, outcome, action taken with IP, and relationship to the IP were listed.
  Non-Treatment-emergent adverse event (non-TEAE): any AE occurring before the first dose of IP, or >30 days after the last dose TEAE: event occurring after first dose of IP or present prior to the first dose, but increasing in severity after IP administration.
Arm/Group | AZD8871 100 µg | AZD8871 600 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/39 | 1/36
Other Adverse Events (participants affected / at risk) | 5/34 | 7/39 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8871 100 µg (N=34) | AZD8871 600 µg (N=39) | Placebo (N=36)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8871 100 µg (N=34) | AZD8871 600 µg (N=39) | Placebo (N=36)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (3) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infections (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and / or presentation whether complete or partial, of any part of the data or results of this study will not be allowed until global publication and study results disclosure by the sponsor as per EMA / FDA regulatory compliance obligations, and only after mutual agreement between the Investigator and AstraZeneca

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT02971293/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02971293/SAP_001.pdf